CLINICAL TRIAL: NCT01474538
Title: A Randomized, Double-Blind, Crossover Trial Comparing the Safety and Efficacy of Insulin Lispro With the Safety and Efficacy of Insulin Aspart in Subjects With Type 2 Diabetes on CSII Therapy
Brief Title: Safety and Efficacy Study of Insulin Lispro Versus Insulin Aspart in Participants With Type 2 Diabetes on Insulin Pump Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 14207; F3Z-MC-IOQH (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Results first posted 2014-03-20 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; type 2 diabetes; insulin pump; continuous subcutaneous insulin infusion; CSII; A1C
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Insulin Lispro; Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Lispro, then Insulin Aspart (Active Comparator): Insulin lispro [100 units/milliliter (U/mL)] administered by continuous subcutaneous insulin infusion (CSII) pump for 16 weeks in Treatment Period 1, followed by insulin aspart (100 U/mL) administered by CSII pump for 16 weeks in Treatment Period 2.
  Interventions: Drug: Insulin Lispro
- Insulin Aspart, then Insulin Lispro (Active Comparator): Insulin aspart (100 U/mL) administered by CSII pump for 16 weeks in Treatment Period 1, followed by insulin lispro (100 U/mL) administered by CSII pump for 16 weeks in Treatment Period 2.
  Interventions: Drug: Insulin Aspart

INTERVENTIONS:
Drug: Insulin Lispro — Insulin lispro (100 U/mL) administered by CSII pump
  Other Names: Humalog; LY275585
  Arms: Insulin Lispro, then Insulin Aspart
Drug: Insulin Aspart — Insulin aspart (100 U/mL) administered by CSII pump
  Other Names: Novolog
  Arms: Insulin Aspart, then Insulin Lispro

SUMMARY:
This study will provide information on the use of insulin lispro and insulin aspart in insulin pumps in participants with type 2 diabetes.

DETAILED DESCRIPTION:
This study will provide clinical information on the use of insulin lispro in continuous subcutaneous insulin infusion (CSII) in participants with type 2 diabetes. This study is designed to allow comparison of the 2 rapid-acting insulin analogs, with regard to their efficacy and safety, when used as a pump insulin therapy in this participant population. Each participant will be randomized to 1 of the 2 sequence groups in a 1:1 ratio and randomization will be stratified according to screening A1C (less than or equal to 8.0% or greater than 8.0%) and thiazolidinedione (TZD) use (yes or no). The study design includes the following periods: Screening/Randomization, Treatment Period 1 (16 weeks), and Treatment Period 2 (16 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes (per World Health Organization [WHO] Classification of Diabetes)
* Have been treated with CSII therapy using a rapid-acting analog for the previous 6 months
* Have a screening A1C less than or equal to 9.0% (no lower limit for A1C)
* Have a body mass index (BMI) less than 45 kilograms/square meter (kg/m²) at screening
* Have a history of stable body weight (not varying by greater than 10% for at least 3 months prior to screening)
* For participants on oral anti-diabetes medications (OAMs): must have been on a stable dose of OAMs, labeled for use with insulin, for at least 3 months prior to study entry

Exclusion Criteria:

* Have severe insulin resistance [require greater than 2 units/kilogram/day (U/kg/day) of insulin]
* Are taking or have taken within the last 3 months, antihyperglycemic medication not approved for use with insulin, injectable non-insulin antihyperglycemic medications, or have a contraindication to current antihyperglycemic medication
* Have a serum creatinine greater than or equal to 2 milligrams/deciliter (mg/dL) if not on metformin; known metabolic or lactic acidosis; any condition associated with hypoperfusion, hypoxemia, dehydration, or sepsis; and/or a radiologic contrast study within 48 hours prior to study entry
* Are receiving chronic (lasting longer than 2 weeks) systemic glucocorticoid therapy (excluding topical, intraocular, intraarticular, and inhaled preparations) or have received such therapy within 2 weeks immediately before screening
* Have had more than 1 episode of hypoglycemia (defined as requiring assistance of a third party due to disabling hypoglycemia) within 6 months prior to entry into the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2011-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-877-615-4559 Mon-Fri 9 AM - 5 PM Eastern Time (UTC/GMT -5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- United States (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metairie, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Asheville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Lispro / Insulin Aspart: Insulin lispro [100 units/milliliter (U/mL)] administered by continuous subcutaneous insulin infusion (CSII) pump for 16 weeks in Treatment Period 1, followed by insulin aspart (100 U/mL) administered by CSII pump for 16 weeks in Treatment Period 2.
- Insulin Aspart / Insulin Lispro: Insulin aspart (100 U/mL) administered by CSII pump for 16 weeks in Treatment Period 1, followed by insulin lispro (100 U/mL) administered by CSII pump for 16 weeks in Treatment Period 2.
Period: Treatment Period 1
Arm/Group | Insulin Lispro / Insulin Aspart | Insulin Aspart / Insulin Lispro
Started | 60 | 62
Received at Least 1 Dose of Study Drug | 60 | 62
Completed | 57 | 58
Not Completed | 3 | 4
Not completed — Death | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Protocol Violation | 0 | 1
Period: Treatment Period 2
Arm/Group | Insulin Lispro / Insulin Aspart | Insulin Aspart / Insulin Lispro
Started | 57 | 58
Received at Least 1 Dose of Study Drug | 57 | 58
Completed | 51 | 56
Not Completed | 6 | 2
Not completed — Death | 1 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Sponsor decision | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Lispro / Insulin Aspart | Insulin Aspart / Insulin Lispro | Total
Number analyzed (Participants) | 60 | 62 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.73 (10.41) | 60.40 (9.72) | 59.58 (10.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 32 | 65
  Male | 27 | 30 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 53 | 54 | 107
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 58 | 61 | 119
Region of Enrollment [Number; unit: participants]
  United States | 60 | 62 | 122

OUTCOME MEASURES:

1. Primary Outcome: Glycosylated Hemoglobin A1C (HbA1c) at Endpoint
Description: Hemoglobin A1c (HbA1c) is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over the last 8-12 weeks. Least Squares (LS) means were adjusted for treatment, period, sequence, thiazolidinedione use (Yes/No), baseline HbA1c (>8% or ≤8%) and participants.
Time Frame: After 16 weeks of each treatment (Periods1 and 2)
Population: All randomized participants who received at least 1 dose of study drug and had HbA1c measured at Week 16 of treatment Period 1 or 2. Participants were analyzed based on the treatment they received.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Groups:
- Insulin Lispro: Insulin lispro [100 units/milliliter (U/mL)] administered by continuous subcutaneous insulin infusion (CSII) pump for 16 weeks in Treatment Period 1 or Treatment Period 2.
- Insulin Aspart: Insulin aspart (100 U/mL) administered by CSII pump for 16 weeks in Treatment Period 1 or Treatment Period 2.
Arm/Group | Insulin Lispro | Insulin Aspart
Number analyzed (Participants) | 112 | 111
percentage of glycosylated hemoglobin | 7.50 (0.12) | 7.40 (0.12)
Statistical Analysis 1: Comparison: Insulin Lispro vs Insulin Aspart; Test type: Non-Inferiority or Equivalence — If the upper limit of the 95% confidence interval (CI) was below 0.4%, lispro was declared non-inferior to aspart; Mixed Models Analysis; LS Mean difference = 0.10, 95% CI 2-sided [-0.002 to 0.210]

2. Secondary Outcome: Total Daily Insulin Dose
Description: Total daily insulin dose was the average of the last 3 days total insulin dose immediately prior to the Week 16 (endpoint) visit of each treatment period. Least Squares (LS) means were adjusted for treatment, period, sequence, thiazolidinedione use (Yes/No), baseline Hemoglobin A1c (HbA1c) (>8% or ≤8%) and participants.
Time Frame: Week 16 of each treatment (Periods 1 and 2)
Population: All randomized participants who received at least 1 dose of study drug and had total daily insulin dose recorded during Treatment Period (TP) 1 or 2. If endpoint data was missing for a specific TP, last observation carried forward (LOCF) method was implemented for that respective TP. Participants were analyzed based on the treatment they received.
Measure: Least Squares Mean (Standard Error); unit: units of insulin
Arm/Group | Insulin Lispro | Insulin Aspart
Number analyzed (Participants) | 116 | 117
units of insulin | 80.41 (4.78) | 80.69 (4.77)
Statistical Analysis 1: Comparison: Insulin Lispro vs Insulin Aspart; Test type: Superiority or Other; Mixed Models Analysis; LS Mean difference = -0.28, 95% CI 2-sided [-2.92 to 2.35]

3. Secondary Outcome: Rate of Hypoglycemic Events Per 30 Days
Description: A hypoglycemic episode is defined as any time a participant feels that he/she is experiencing a sign or symptom that is associated with hypoglycemia, or has blood glucose concentration of ≤70 milligrams/deciliter [mg/dL (3.9 millimoles/liter (mmol/L)]. Least Squares (LS) means were adjusted for treatment, period, sequence, baseline hypoglycemic event rate, thiazolidinedione use (Yes/No) and baseline Hemoglobin A1c (HbA1c) (>8% or ≤8%).
Time Frame: Baseline through 16 weeks of each treatment (Periods 1 and 2)
Population: All randomized participants who received at least 1 dose of study drug. Participants were analyzed based on the treatment they received.
Measure: Least Squares Mean (Standard Error); unit: hypoglycemic events per 30 days
Arm/Group | Insulin Lispro | Insulin Aspart
Number analyzed (Participants) | 118 | 119
hypoglycemic events per 30 days | 2.24 (0.28) | 2.38 (0.29)
Statistical Analysis 1: Comparison: Insulin Lispro vs Insulin Aspart; Test type: Superiority or Other; p = 0.522, Negative binomial; LS Mean Ratio = 0.94

4. Secondary Outcome: Change From Baseline in Weight
Description: Least Squares (LS) means were adjusted for treatment, period, sequence, thiazolidinedione use (Yes/No), baseline Hemoglobin A1c (HbA1c) (>8% or ≤8%), baseline weight and participants.
Time Frame: Baseline, Week 16 of treatment Periods 1 and 2
Population: All randomized participants who received at least 1 dose of study drug and had weight measured at baseline and Week 16 of Treatment Period 1 or 2. Participants were analyzed based on the treatment they received.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | Insulin Lispro | Insulin Aspart
Number analyzed (Participants) | 116 | 117
kilograms (kg) | 0.31 (0.53) | 0.89 (0.52)
Statistical Analysis 1: Comparison: Insulin Lispro vs Insulin Aspart; Test type: Superiority or Other; p = 0.216, Grizzle Model; LS Mean difference = -0.58

5. Secondary Outcome: Percentage of Participants With Hypoglycemic Events
Description: A hypoglycemic episode is defined as any time a participant feels that he/she is experiencing a sign or symptom that is associated with hypoglycemia, or has blood glucose concentration of ≤ 70 milligrams/deciliter [mg/dL (3.9 millimoles/liter (mmol/L)]. The percentage of participants is the total number of participants experiencing hypoglycemic events divided by number of participants in the treatment arm multiplied by 100.
Time Frame: Baseline through 16 weeks of each treatment (Periods 1 and 2)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Lispro | Insulin Aspart
Number analyzed (Participants) | 118 | 119
percentage of participants | 71.2 | 74.8
Statistical Analysis 1: Comparison: Insulin Lispro vs Insulin Aspart; Test type: Superiority or Other; p = 0.471, Prescott test

ADVERSE EVENTS:
Arm/Group | Insulin Lispro | Insulin Aspart
Serious Adverse Events (participants affected / at risk) | 15/118 | 14/119
Other Adverse Events (participants affected / at risk) | 59/118 | 62/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Insulin Lispro (N=118) | Insulin Aspart (N=119)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 3 (3) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) — Event resulted in death in Insulin Aspart group.
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Infusion site abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Event resulted in death.
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
International normalised ratio decreased (Investigations) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 0/55 (0) | 1/55 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Insulin Lispro (N=118) | Insulin Aspart (N=119)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 2 (2)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Iritis (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Parotid gland inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (4) | 4 (4)
Injection site haematoma (General disorders) | 1 (1) | 0 (0)
Injection site nodule (General disorders) | 2 (2) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Oedema (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Multiple allergies (Immune system disorders) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 1 (2)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 2 (2)
Infusion site infection (Infections and infestations) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (5) | 5 (6)
Onychomycosis (Infections and infestations) | 1 (1) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 4 (4)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Angiogram peripheral (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Catheterisation cardiac (Investigations) | 0 (0) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 2 (2) | 2 (2)
International normalised ratio decreased (Investigations) | 1 (1) | 1 (1)
Pulse pressure decreased (Investigations) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Bunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Essential tremor (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1/63 (1) | 1/64 (2)
Prostatitis (Reproductive system and breast disorders) | 1/55 (1) | 0/55 (0)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 0/63 (0) | 1/64 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Arterial repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Foraminotomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastric banding (Surgical and medical procedures) | 0 (0) | 1 (1)
Mole excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Rotator cuff repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal fusion surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal laminectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Angiopathy (Vascular disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 2 (2)
Intermittent claudication (Vascular disorders) | 1 (1) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days